CLINICAL TRIAL: NCT01681082
Title: Psychological Effects of Tai Chi Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SE-2012-0539
Record Dates: First submitted 2012-08-30; First posted 2012-09-07 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2015-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

ARMS (2):
- Tai Chi Training (Experimental): Subjects will be recruited from the University of Wisconsin-Madison course, "Introduction to Martial Arts: Tai Chi".
  Interventions: Behavioral: Tai Chi training
- Control (No Intervention): Subjects will be recruited from the University of Wisconsin-Madison course "Introduction to Psychology".

INTERVENTIONS:
Behavioral: Tai Chi training — 24 form Yang style Tai Chi. 50 minute sessions, twice weekly.
  Arms: Tai Chi Training

SUMMARY:
The general purpose of this study is to examine the effect of tai chi training on cognitive function in young adults. The investigators will test subjects enrolled in a semester-long tai chi course along with control subjects. The specific aims are to measure duration of practice, cognitive function, physical balance, and Attention Deficit Hyperactivity Disorder (ADHD) indicators. The investigators primary hypotheses are that, compared to controls, subjects in the tai chi course will show improvements in (1a) spatial working memory and (1b) response inhibition. The investigators secondary hypotheses are that, among the subjects participating in the tai chi course, these cognitive improvements will correlate with (2a) improvements in balance and (2b) duration of tai chi practice, and that, among all participants, (2c) ADHD indications will correlate with cognitive measures.

ELIGIBILITY:
Inclusion Criteria:

* Able to perform balance and cognitive tests

Exclusion Criteria:

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in working memory | Baseline and 14 weeks
  CANTAB Spatial Working Memory Task: SWM between errors

SECONDARY OUTCOMES:
Change in physical balance | Baseline and 14 weeks
  One Legged Stance Test. Time standing on one leg with eyes closed. Average over left and right leg of best of three trials on each side.
Change in impulsivity | Baseline and 14 weeks
  CANTAB Stop Signal Task: reaction time (SSRT).
Change in affective processing | Baseline and 14 weeks
  CANTAB Affective Go/No-Go Task: mean correct latency
Change in attention deficit hyperactivity disorder (ADHD) scale | Baseline and 14 weeks
  World Health Organization adult ADHD self-report scale (ASRS). Scoring of 6 item ASRS screener per Kessler et al. Psychological Medicine (2005) 35:245-256.
Duration of practice | 14 weeks
  Total minutes of tai chi practice including class time.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander K. Converse, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Waisman Center, Madison, Wisconsin, United States

REFERENCES:
- [Result] Converse AK, Ahlers EO, Travers BG, Davidson RJ. Tai chi training reduces self-report of inattention in healthy young adults. Front Hum Neurosci. 2014 Jan 27;8:13. doi: 10.3389/fnhum.2014.00013. eCollection 2014. PMID 24478679